CLINICAL TRIAL: NCT05435781
Title: RESCUE - Effect of Supplemental Hydrocortisone During Stress in Prednisolone-induced Adrenal Insufficiency; A Multicentre, Randomised, Double Blinded, Placebo-controlled Clinical Trial on Health-related Quality of Life in Patients With Polymyalgia Rheumatica/Giant Cell Arteritis Receiving Ongoing Low-dose Prednisolone Treatment.
Brief Title: Effect of Supplemental Hydrocortisone During Stress in Prednisolone-induced Adrenal Insufficiency
Acronym: RESCUE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ulla Feldt-Rasmussen (Other)
Collaborators: Aarhus University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Sponsor-Investigator, Ulla Feldt-Rasmussen, Professor, Senior Consultant Ulla Feldt-Rasmussen, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RESCUE; 2021-002528-18 (EudraCT Number); H-21041930 (Other: The Committees of Health Research Ethics in the Capital Region of Denmark)
Record Dates: First submitted 2022-06-13; First posted 2022-06-28 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Adrenal Insufficiency; Polymyalgia Rheumatica; Giant Cell Arteritis
Keywords: Glucocorticoid-induced adrenal insufficiency; Prednisolone; Glucocorticoids; Hypothalamic-pituitary-adrenal axis
MeSH Terms: conditions — Adrenal Insufficiency; Polymyalgia Rheumatica; Giant Cell Arteritis | interventions — Hydrocortisone

STUDY DESIGN:
Intervention Model Description: Double-blinded randomised placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients and all study personnel are blinded for study medication (hydrocortisone or placebo)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- RCT group - hydrocortisone (Active Comparator): Patients with polymyalgia rheumatica/giant cell arteritis with glucocorticoid-induced adrenal insufficiency (Synacthen test response <420 nmol/l) that are randomised to receive hydrocortisone
  Interventions: Drug: Hydrocortisone
- RCT group - placebo (Placebo Comparator): Patients with polymyalgia rheumatica/giant cell arteritis with glucocorticoid-induced adrenal insufficiency (Synacthen test response <420 nmol/l) that are randomised to receive placebo
  Interventions: Drug: Placebo for hydrocortisone
- Control group (No Intervention): Patients with polymyalgia rheumatica/giant cell arteritis with normal adrenal function (Synacthen test response ≥420 nmol/l)

INTERVENTIONS:
Drug: Hydrocortisone — Patients are randomised to either placebo or hydrocortisone supplemental doses in situations of stress. Patients will continue prednisolone treatment and tapering hereof according to current clinical guidelines for PMR/GCA , prednisolone is not part of the intervention.
  Arms: RCT group - hydrocortisone
Drug: Placebo for hydrocortisone — Patients are randomised to either placebo or hydrocortisone supplemental doses in situations of stress. Patients will continue prednisolone treatment and tapering hereof according to current clinical guidelines for PMR/GCA , prednisolone is not part of the intervention.
  Arms: RCT group - placebo

SUMMARY:
In this double-blinded randomised placebo-controlled clinical trial, the aim is to determine the effect of supplemental hydrocortisone compared with placebo during mild to moderate physical or mental stress on health related quality of life in patients with polymyalgia rheumatica (PMR)/giant cell arteritis (GCA) on ongoing low-dose prednisolone diagnosed with glucocorticoid-induced adrenal insufficiency. The main emphasis is on fatigue (primary outcome) and daily variation hereof during periods of stress.

DETAILED DESCRIPTION:
The study will include patients with PMR/GCA on ongoing prednisolone treatment in a low dose of > 0 mg/day and ≤5mg/day. Eligible patients will undergo a Synacthen® test and 250 patients with a stimulated cortisol level <420 nmol/l (biochemical adrenal insufficiency) will be randomised to either placebo or hydrocortisone supplemental doses during stress. Patients will continue prednisolone treatment and tapering hereof according to current clinical guidelines for PMR/GCA and add supplemental hydrocortisone/placebo in situations of stress according to study protocol. In situations of severe stress (potential adrenal crisis) patients will receive open label hydrocortisone treatment according to routine clinical care. The duration of RESCUE is 6 months but stops earlier if the patient stops prednisolone treatment earlier. In case of a flare of PMR/GCA during the study where prednisolone is increased to >5mg/day for e.g. 5 weeks the study is prolonged accordingly 5 weeks.

Seventy-five patients with stimulated cortisol ≥420 nmol/l (normal adrenal function) will be used as a reference group. The participants will undergo screening and baseline examinations, 3 month's reporting of HRQoL, and with patient consent follow-up through medical records on prednisolone treatment characteristics, and number of hospitalisations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Women must be postmenopausal (FSH is measured at the screening visit)
* A diagnosis of PMR/GCA, or both conditions combined.
* Treatment with prednisolone ≥12 weeks
* Ongoing prednisolone treatment, with current daily prednisolone dose > 0 mg and ≤5 mg. The dose must have been ≤5 mg for minimum 2 weeks at the time of the screening visit.

Exclusion Criteria:

* Known primary or secondary adrenal insufficiency
* Known Cushing's Syndrome
* Known allergy towards study medication ingredients
* Severe comorbidity: Heart failure (New York Heart Association class IV); Kidney failure with an estimated glomerular filtration rate <30 mL/min (Chronic kidney disease stage 4-5); Liver disease in the form of cirrhosis; Active cancer; Known severe immune deficiency; A history of psychiatric disease requiring treatment by a psychiatric department (for affective disorders only if within the last year before study entry)
* Alcohol consumption >21 units per week
* Planned major surgery during the study period at study entry.
* Use of drugs that interfere with cortisol metabolism/measurements: Systemic oestrogen treatment (discontinued < 1 month before inclusion), Treatment with strong CYP3A4 inhibitors or inducers, Use of other glucocorticoid formulations (Inhaled corticosteroids, intraarticular or intramuscular injections, steroid creams European steroid group IV-V used in the genital area. Note: Permitted glucocorticoid formulations: Eye-drops, nasal spray, glucocorticoid creams European steroid group I-III, and European steroid group IV-V used in the non-genital area only.)
* Inability to provide written informed consent.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
ecological momentary assessments (EMA) of the Multidimensional Fatigue Inventory (MFI-20) General Fatigue scale, adjusted for EMA | In situations of stress, participants are asked to answer the EMA items 5 times daily at semi-randomised time points, for 3 days. Diurnal profiles are generated and one diurnal profile summarizes responses during the day across all 'sick-days'.
  EMA in situations of stress. EMA reporting will be conducted electronically on a smartphone.

SECONDARY OUTCOMES:
Daily 'end-of-day' app-facilitated patient reported outcome (PRO) assessments | Patients are asked daily throughout the study period as 'end-of-day' assessments.
  Key secondary outcome - obtain information about intercurrent illness, injury, or stress, and symptoms of fatigue, nausea, and general malaise. The questions about symptoms originate from the Danish version of the PRO-CTCAE.
SF-36 | At baseline, 3 months and 6 months
  Key secondary outcome
AddiQol-30 | At baseline, 3 months and 6 months
  Key secondary outcome
PMR/GCA treatment characteristics -accumulated glucocorticoid dose | Information from 6 months before baseline to end-of study
  Key secondary outcome. accumulated glucocorticoid dose
PMR/GCA treatment characteristics -prednisolone treatment duration | Information from 6 months before baseline to end-of study
  Key secondary outcome. Duration of prednisolone treatment, duration of prednisolone tapering (5 mg - 0 mg)
Number of 'sick days' | Throughout study period (6 months)
  Key secondary outcome
Incidens of adrenal crises and hospitalisations | Throughout study period (6 months)
  Incidence rate of adrenal crises and hospitalisations
Adrenal crises grading | Throughout study period (6 months)
  Grade of adrenal crises.
Body composition and muscle strength - DXA scan | Baseline and 6 months
  Safety outcome for exogenous Cushing's Syndrome (Dual-energy X-ray absorptiometry (DXA) scan: fat percentage, body composition
Body composition and muscle strength - Waist, hip, height | Baseline and 6 months
  Safety outcome for exogenous Cushing's Syndrome (Waist, hip, height)
Body composition and muscle strength -weight | Baseline and 6 months
  Safety outcome for exogenous Cushing's Syndrome (weight)
Body composition and muscle strength - body mass index (BMI) | Baseline and 6 months
  Safety outcome for exogenous Cushing's Syndrome (BMI)
Body composition and muscle strength - Timed up and go | Baseline and 6 months
  Safety outcome for exogenous Cushing's Syndrome (Timed up and go)
Body composition and muscle strength - Handgrip strength | Baseline and 6 months
  Safety outcome for exogenous Cushing's Syndrome (Handgrip strength)
Body composition and muscle strength - Short Physical Performance Battery | Baseline and 6 months
  Safety outcome for exogenous Cushing's Syndrome (Short Physical Performance Battery)
Body composition and muscle strength - Chair rising test | Baseline and 6 months
  Safety outcome for exogenous Cushing's Syndrome (Chair rising test)
Bone quality - Dual-energy X-ray absorptiometry (DXA) scan | Baseline and 6 months
  Safety outcome for exogenous Cushing's Syndrome (DXA scan, vertebral and hip)
Bone quality - bone markers in blood and urine | Baseline and 6 months
  Safety outcome for exogenous Cushing's Syndrome (bone markers in blood and urine)
Metabolic and cardiovascular risk - Automated office blood pressure | Baseline and 6 months
  Safety outcome for exogenous Cushing's Syndrome (Automated office blood pressure)
Metabolic and cardiovascular risk (Coagulation and Inflammation markers in blood) | Baseline and 6 months
  Safety outcome for exogenous Cushing's Syndrome (Coagulation and Inflammation markers in blood)
Metabolic and cardiovascular risk - Metabolic and cardiovascular markers in blood and urine | Baseline and 6 months
  Safety outcome for exogenous Cushing's Syndrome (Metabolic and cardiovascular markers in blood and urine)
Patient reported symptoms of hypercortisolism - CushingQol | Baseline and 6 months
  Safety outcome for exogenous Cushing's Syndrome (CushingQol)
Patient reported symptoms of hypercortisolism - Single item Sleep Quality Scale (SQS)) | Baseline and 6 months
  Safety outcome for exogenous Cushing's Syndrome (Single item Sleep Quality Scale (SQS))
Biological integrated cortisol status assessment - ACTH test | At baseline, (3 months) and 6 months
  ACTH test for normalization of adrenal function
Biological integrated cortisol status assessment - 24h urine | At baseline, (3 months) and 6 months
  24h urine for cortisol and metabolites.
Biological integrated cortisol status assessment - Salivary cortisol/cortisone | At baseline, (3 months) and 6 months
  Salivary cortisol/cortisone
Biological integrated cortisol status assessment - Circulating biomarkers of glucocorticoid effects and adverse effects | At baseline, (3 months) and 6 months
  Circulating biomarkers of glucocorticoid effects and adverse effects.
Biological integrated cortisol status assessment - P-cortisol after 24 hours prednisolone pause. | At baseline, (3 months) and 6 months
  P-cortisol after 24 hours prednisolone pause.
ecological momentary assessments (EMA) of the Multidimensional Fatigue Inventory (MFI-20) General Fatigue scale, adjusted for EMA | EMA is used at fixed time points monthly. Participants are asked to answer the EMA items 5 times daily at semi-randomised time points, for 3 days. Diurnal profiles are generated and one diurnal profile summarizes responses during the day across all days.
  EMA in situations without stress, key-secondary putcome: EMA reporting will be conducted electronically on a smartphone

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Feldt-Rasmussen, Professor, Principal Investigator — Rigshospitalet, Denmark
Locations (3):
- Denmark (3):
  - Department of Endocrinology, Aarhus University Hospital, Aarhus
  - Department of Medical Endocrinology, Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Department of Endocrinology, Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No